CLINICAL TRIAL: NCT05504369
Title: Effects of Magnetic Tape on the Autonomic Nervous System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida Gulf Coast University (Other)
Collaborators: University of Valencia (Other)
Responsible Party: Principal Investigator, Dr. Rob Sillevis,, Associate Professor, Florida Gulf Coast University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: 1240878
Record Dates: First submitted 2022-08-10; First posted 2022-08-17 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Low Back Pain
Keywords: Magnetic tape; magnetic nano particles; Pupillometry; Autonomic nervous system; lower back pain; PA test; Skin pinch test
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: Single group design with random allocation of intervention placebo versus treatment tape. Next day other intervention was used
Who Masked: Participant, Investigator
Masking Description: Participant and researchers where not aware of the magnetic tape versus placebo tape as the look and feel identical
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Magnetic tape arm (Active Comparator): Tape application bilaterally in the lumbar spine
  Interventions: Other: Magnetic tape
- Placebo tape arm (Sham Comparator): Tape application bilaterally in the lumbar spine
  Interventions: Other: Placebo tape

INTERVENTIONS:
Other: Magnetic tape — Tape with magnetic nanoparticles applied to the skin
  Arms: Magnetic tape arm
Other: Placebo tape — Tape without nano particles applied to the skin
  Arms: Placebo tape arm

SUMMARY:
The effect of magnetic tape on pain and autonomic nervous system in subject with lower back pain.

DETAILED DESCRIPTION:
The effects of magnetic nanoparticles in tape applied in the lumbar spine on the autonomic nervous system measured with fully automated pupillometry and on pain in the spine measured with posterior to anterior pressure on the spinous process and the skin pinch test paravertebrally

ELIGIBILITY:
Inclusion Criteria:

* Current lower back pain with NPRS of 5
* Between ages 18-65

Exclusion Criteria:

* No lower back pain or pain <5 on the NPRS
* Not meeting age limit
* Having condition that prevents the PA procedure
* Conditions of the nervous system and inability keep eyes open

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Pupillometry | 60 seconds measure preceding tape application. After outcome 5
  1 minute continues pupil diameter measure
Pupillometry | Second 60 second measure immediate after tape application. After outcome 1
  1 minute continues pupil diameter measure
Pupillometry | Third 60 measure 3 minutes after the tape is removed. After outcome 2
  1 minute continues pupil diameter measure

SECONDARY OUTCOMES:
PA spine | First PA measure of 5 seconds on each PA of 5 seconds on each segment is starting off the measurement phase. This is the first outcome measure
  Anterior (PA) pressure on each spinal segment
Skin pinch test | 3 seconds skin pinch test at each level starting immediately following the first PA measure. After Outcome 4
  Bilaterally of each vertebrae
PA spine | Five second measure of PA of 5 seconds each segment is taken immediately after the third pupillometry measure (tape removed). After outcome 3
  Anterior (PA) pressure on each spinal segment
Skin Pinch test | 3 seconds skin pinch test at each level starting immediately following outcome 6
  Bilaterally of each vertebrae

CONTACTS AND LOCATIONS:
Locations (1):
- University of Valencia, Valencia de Alcántara, Spain

IPD SHARING:
Plan to Share IPD: No
No plan in place